CLINICAL TRIAL: NCT05115175
Title: Mindfulness and Diabetes Distress: Acceptability of Self-Led Mindfulness-Based Intervention
Brief Title: Acceptability of Self-Led Mindfulness-Based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Collaborators: AlterMed Research foundation (Unknown)
Responsible Party: Principal Investigator, Holly Hazlett-Stevens, Associate Professor, University of Nevada, Reno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1221205
Record Dates: First submitted 2021-10-11; First posted 2021-11-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes distress; adolescents; mindfulness; psychosocial intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Adolescents (N=25) aged 14 to 18 diagnosed with type 1 diabetes completed a baseline assessment. Participants were randomized to receive a 10-week self-guided mindfulness-based stress reduction program immediately (n=10) or after a 10-week wait (n=15). During the intervention period, participants completed weekly assignments and qualitative and quantitative feedback surveys. At 10-weeks and 20-weeks follow-up assessments were completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention immediately (Experimental): The intervention was delivered via a teen MBSR workbook and online communication across the 10-week intervention period. Participants were assigned weekly readings and activities from an MBSR workbook for teens. Topics included understanding stress, introduction to mindfulness, mindful eating and other mindfulness-based intervention principles and were recommended to be completed daily. Mindfulness-based exercises were either self-led per instructions provided in the workbook or to be completed using an audio recording directing participants' behaviors during the exercise.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Intervention in ten weeks following waitlist (Experimental): This group received the same intervention as the first arm, however, the participants in arm 2 received the intervention after a 10-week waitlist period. The intervention was delivered via a teen MBSR workbook and online communication across the 10-week intervention period. Participants were assigned weekly readings and activities from an MBSR workbook for teens. Topics included understanding stress, introduction to mindfulness, mindful eating and other mindfulness-based intervention principles and were recommended to be completed daily. Mindfulness-based exercises were either self-led per instructions provided in the workbook or to be completed using an audio recording directing participants' behaviors during the exercise.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — Participants engaged in meditation and self-led exercises to help them understand and cope with stress.

SUMMARY:
This study had two primary aims. First, the investigators examined the associations between mindfulness and diabetes-related outcomes. It was hypothesized that at baseline, increased mindfulness would be associated with decreased diabetes distress and more optimal glycemic levels and that all three variables would share similar associations with related constructs including greater self-compassion, lower general stress, better psychosocial health, increased diabetes treatment engagement, and greater diabetes-related quality of life. The association between specific aspects of dispositional mindfulness and diabetes distress was also explored. Second, the investigators examined the acceptability, feasibility, and potential utility of self-led MBSR intervention. It was hypothesized that participation in a self-led MBSR intervention would be feasible and acceptable, evidenced by treatment attrition and participant feedback. It was also hypothesized that participants who received the self-led Mindfulness-based stress reduction (MBSR) intervention would experience increased mindfulness and decreased diabetes distress compared to a waitlist control group.

DETAILED DESCRIPTION:
The goal of the present study was to assess the associations of dispositional mindfulness, diabetes distress, and glycemic outcomes for adolescents with type 1 diabetes as well as to use an iterative approach to developing a self-led scalable mindfulness-based intervention. A self-led mindfulness-based intervention may provide a mindfulness practice to help adolescents with type 1 diabetes improve glycemic outcomes through diabetes distress reduction while also being practical within a pediatric endocrinology clinic. A self-led intervention may also reduce the burden associated with mindfulness-based interventions. This is important considering the heightened emotional and time burden adolescents may already experience due to disease management and the intensity of a traditional mindfulness-based intervention.

This study had two primary aims. First, the investigators examined the associations between mindfulness and diabetes-related outcomes. It was hypothesized that at baseline, increased mindfulness would be associated with decreased diabetes distress and more optimal glycemic levels and that all three variables would share similar associations with related constructs including greater self-compassion, lower general stress, better psychosocial health, increased diabetes treatment engagement, and greater diabetes-related quality of life. The association between specific aspects of dispositional mindfulness and diabetes distress was also explored. Second, the investigators examined the acceptability, feasibility, and potential utility of self-led MBSR intervention. It was hypothesized that participation in a self-led MBSR intervention would be feasible and acceptable, evidenced by treatment attrition and participant feedback. It was also hypothesized that participants who received the self-led MBSR intervention would experience increased mindfulness and decreased diabetes distress compared to a waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-19 years old
* Type 1 diabetes diagnosis
* Currently attending school or a recent high school graduate

Exclusion Criteria:

* Ward of the state
* Severe psychiatric disturbances (e.g., active psychosis)
* Severe developmental delay that hindered ability to self-report

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Mindfulness as Assessed by Mindful Attention Awareness Scale-Adolescent (MAAS-A) | 10 weeks intervention, 20 weeks waitlist
  Assessed difference in dispositional mindfulness in adolescents from pre-intervention to post-intervention. The Mindful Attention Awareness Scale-Adolescent has a single-factor structure with 14 items rated on a 6-point scale (1 = almost always, 6 = almost never). Higher scores indicate higher trait mindfulness.
Change from Baseline in Engagement in Self-Compassionate Behavior as Assessed by Self-Compassion Scale (SCS) | 10 weeks intervention, 20 weeks waitlist
  Participants rated how often they engage in each self-compassionate behavior in specific situations pre- and post-intervention. The Self-Compassion Scale is a 26-item measure rated on a 5-point scale (1 = almost never, 5 = almost always). Higher scores indicate higher self-compassion.
Change from Baseline in Diabetes Stress as Assessed by Diabetes Stress Questionnaire (DSQ) | 10 weeks intervention, 20 weeks waitlist
  Assessed different daily, diabetes-specific stressors from pre-intervention to post-intervention. The Diabetes Stress Questionnaire consists of 65 items and includes eight subscales. Participants rate severity of stress across several diabetes-related scenarios on a 4-point scale (0 = not at all, 3 = very much). Higher scores indicate higher diabetes distress.
Change from Baseline in Health-Related Quality of Life as Assessed by Pediatric Quality of Life Inventory (PedsQL) 3.2 Diabetes Module | 10 weeks intervention, 20 weeks waitlist
  Assessed diabetes-specific, health-related quality of life in children, adolescents, and young adults from pre-intervention to post-intervention. The Pediatric Quality of Life Inventory 3.2 Diabetes Module consists of 33 items rated on a 5-point scale (0 = never, 4 = almost always). Higher scores indicate greater quality of life.
Change from Baseline in Perceived Stress as Assessed by Perceived Stress Scale-10 Item Version (PSS-10) | 10 weeks intervention, 20 weeks waitlist
  Assessed the severity of broad, stressful situations in adolescents from pre-intervention to post-intervention. Participants rank how often each statement applies to their feelings of stress on a 5-point scale (0 = never, 4 = very often). Negative items are reversed and the sum of all 10 items is calculated. Higher scores indicate higher perceived stress.
Change from Baseline in Psychosocial Impairment as Assessed by Pediatric Symptoms Checklist-17 (PSC-17) | 10 weeks intervention, 20 weeks waitlist
  Assessed psychosocial functioning from pre-intervention to post-intervention. Participants rate how frequently each symptom occurs on a 3-point scale (0 = never, 2 = often). Total scores range from 0-34 with higher scores indicating greater risk of psychosocial impairment.
Change from Baseline in Diabetes Treatment Engagement as Assessed by Self Care Inventory (SCI) | 10 weeks intervention, 20 weeks waitlist
  Assessed to what degree individuals follow health care provider guidelines for diabetes-management behaviors from pre-intervention to post-intervention. The investigators removed the item "how frequently do you come in for appointments" from the study as the measure was not used within a physician/ appointment context. After removing the item, the Self Care Inventory consisted of 22 items and is rated on a 5-point scale (1 = never, 5 = always). Higher scores indicate higher diabetes treatment engagement.
Change from Baseline in Glycosylated Hemoglobin Percentage | 10 weeks intervention, 20 weeks waitlist
  Assessed the difference in glycosylated hemoglobin percentage from pre-intervention to post-intervention.
Engagement with the Scaled Mindfulness-Based Intervention as Assessed by Number of Weekly Surveys Completed. | 20 weeks
  Assessed the number of weekly surveys each participant completed during the intervention period. Participants were asked to complete at least 6 out of the 10 weekly surveys during the intervention period to be considered highly engaged.
Feasibility of the Scaled Mindfulness-Based Intervention as Assessed by Participant Feedback | 20 weeks
  Assessed the acceptability and feasibility of a mindfulness-based intervention for teens with type 1 diabetes by examining participant feedback on reasons for attrition and low engagement. Weekly feedback surveys asked about barriers to engaging in the weekly material.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Hazlett-Stevens, Ph.D., Principal Investigator — University of Nevada, Reno; Amy Hughes Lansing, Ph.D., Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Overall analyses and scales can be shared as described in participant consent, however, individual participant data will not be shared.

REFERENCES:
- [Background] Shubrook JH, Brannan GD, Wapner A, Klein G, Schwartz FL. Time Needed for Diabetes Self-Care: Nationwide Survey of Certified Diabetes Educators. Diabetes Spectr. 2018 Aug;31(3):267-271. doi: 10.2337/ds17-0077. PMID 30140143
- [Background] Brown KW, West AM, Loverich TM, Biegel GM. Assessing adolescent mindfulness: validation of an adapted Mindful Attention Awareness Scale in adolescent normative and psychiatric populations. Psychol Assess. 2011 Dec;23(4):1023-33. doi: 10.1037/a0021338. Epub 2011 Feb 14. PMID 21319908
- [Background] Neff KD, Bluth K, Toth-Kiraly I, Davidson O, Knox MC, Williamson Z, Costigan A. Development and Validation of the Self-Compassion Scale for Youth. J Pers Assess. 2021 Jan-Feb;103(1):92-105. doi: 10.1080/00223891.2020.1729774. Epub 2020 Mar 3. PMID 32125190
- [Background] Delamater AM, Patino-Fernandez AM, Smith KE, Bubb J. Measurement of diabetes stress in older children and adolescents with type 1 diabetes mellitus. Pediatr Diabetes. 2013 Feb;14(1):50-6. doi: 10.1111/j.1399-5448.2012.00894.x. Epub 2012 Aug 23. PMID 22913570
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Varni JW, Delamater AM, Hood KK, Raymond JK, Chang NT, Driscoll KA, Wong JC, Yi-Frazier JP, Grishman EK, Faith MA, Corathers SD, Kichler JC, Miller JL, Doskey EM, Heffer RW, Wilson DP; Pediatric Quality of Life Inventory 3.2 Diabetes Module Testing Study Consortium. PedsQL 3.2 Diabetes Module for Children, Adolescents, and Young Adults: Reliability and Validity in Type 1 Diabetes. Diabetes Care. 2018 Oct;41(10):2064-2071. doi: 10.2337/dc17-2707. Epub 2018 Jul 30. PMID 30061317
- [Background] Gardner, W., Murphy, M., Childs, G., Kelleher, K., Pagano, M., Jellinek, M., ... & Chiappetta, L. (1999). The PSC-17: A brief pediatric symptom checklist with psychosocial problem subscales. A report from PROS and ASPN. Ambulatory Child Health, 5, 225-225.
- [Background] La Greca, A., Swales, T., Klemp, S., & Madigan, S. (1988). Self-care behaviors among adolescents with diabetes. Proceedings of the Ninth Annual Sessions of the Society of Behavioral Medicine.
- [Derived] Humiston T, Cummings C, Suss S, Cohen LB, Hazlett-Stevens H, Hughes Lansing A. Acceptability of a Self-Led Mindfulness-Based Intervention for Teens with Type 1 Diabetes: Pilot Randomized Controlled Trial. JMIR Form Res. 2024 Jan 30;8:e45659. doi: 10.2196/45659. PMID 38289663

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT05115175/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT05115175/ICF_001.pdf